CLINICAL TRIAL: NCT00028704
Title: Conservative Local Treatment Versus Mastectomy After Induction Chemotherapy In Locally Advanced Breast Cancer: A Randomized Phase III Study
Brief Title: Breast-Conserving Therapy Compared With Mastectomy Followed By Radiation Therapy in Treating Women With Locally Advanced Breast Cancer Previously Treated With Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Central and Eastern European Oncology Group (Other); Grupo Oncologico Cooperativo Chileno de Investigation (Network); International Collaborative Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-10974-22002; EORTC-10974; CEEOG-EORTC-10974; EORTC-22002; GOCCHI-EORTC-10974; ICCG-EORTC-10974; EORTC-BIG-0002; LAMANOMA
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Breast-conserving treatments such as radiation therapy or limited surgery are less invasive than mastectomy and may improve the quality of life. It is not yet known if breast-conserving treatments are as effective as mastectomy followed by radiation therapy in treating locally advanced breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of breast-conserving therapy with mastectomy followed by radiation therapy in treating women who have locally advanced breast cancer that has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and time to loco-regional failure in women with locally advanced breast cancer treated with breast-conserving local therapy vs mastectomy followed by radiotherapy after they have received prior induction chemotherapy.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, initial stage (T0, T1, T2, T3, or Tx vs T4), response to prior induction chemotherapy (complete response (CR) vs other), and menopausal status (premenopausal vs postmenopausal). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo mastectomy followed by radiotherapy.
* Arm II: Patients receive breast-conserving treatment comprising 1 of 3 of the following therapeutic options:

  * Regimen A: Patients receive radiotherapy alone.
  * Regimen B: Patients with a partial response (PR) to prior induction chemotherapy undergo limited surgery followed by radiotherapy. Patients with a CR to prior induction chemotherapy undergo radiotherapy alone.
  * Regimen C: Patients with a partial response (PR) or CR to prior induction chemotherapy undergo radiotherapy alone.

Patients with a CR to radiotherapy receive no further treatment. Patients with a PR to radiotherapy undergo limited surgery.

Quality of life is assessed at baseline, at the end of therapy, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

Patients are followed within 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,300 patients (650 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced breast cancer

  * T3 inoperable, N0-N2
  * Any T, N2
  * T4, N0-N2
  * Inflammatory breast carcinoma
* Prior treatment with 4-6 courses of standard induction chemotherapy or active investigational regimens completed within the past 4 weeks
* Residual tumor size less than 5 cm
* No fixed axillary lymph nodes
* No multifocal or bilateral breast cancer
* No clinical suspicion of extensive ductal carcinoma in situ
* No unresolved skin edema
* No distant metastases (including ipsilateral supraclavicular node)

  * Positive bone scan allowed provided there are no bone metastases on x-ray
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT and SGPT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal:

* Creatinine less than 1.5 times normal

Other:

* No other prior or concurrent malignancy except adequately treated squamous cell or basal cell skin cancer or adequately treated cone-biopsied carcinoma in situ of the cervix
* No serious underlying medical illness that would preclude study
* No psychiatric or addictive disorder that would preclude study
* No contraindication to study treatment
* Not pregnant
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* No concurrent hormonal replacement therapy
* No concurrent oral contraceptives

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for breast cancer

Surgery:

* No prior surgery for breast cancer other than biopsy for diagnosis confirmation

Other:

* No other prior systemic therapy for breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-10; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Jassem, MD, PhD, Study Chair — Medical University of Gdansk; G. van Tienhoven, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marzena Welnicka-Jaskiewicz, MD, Study Chair — Medical University of Gdansk; Rodrigo Arriagada, MD, Study Chair — Instituto de Radiomedicina; Marie Emson, BSc, Study Chair — International Collaborative Cancer Group
Locations (13):
- Belgium (2):
  - Centre Hospitalier Etterbeek Ixelles, Brussels
  - U.Z. Gasthuisberg, Leuven
- Instituto de Radiomedicina, Santiago, Chile
- Rambam Medical Center, Haifa, Israel
- Netherlands (4):
  - Akademisch Medisch Centrum, Amsterdam
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Leiden University Medical Center, Leiden
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Poland (3):
  - Medical University of Gdansk, Gdansk
  - Karol Marcinkowski University, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Charing Cross Hospital, London, England, United Kingdom

REFERENCES:
- [Result] Sinacki M, Jassem J, van Tienhoven G. Conservative local treatment versus mastectomy after induction chemotherapy in locally advanced breast cancer: a randomised phase III study (EORTC 10974/22002, LAMANOMA)--why did this study fail? Eur J Cancer. 2005 Dec;41(18):2787-8. doi: 10.1016/j.ejca.2005.06.027. Epub 2005 Nov 7. No abstract available. PMID 16274985